CLINICAL TRIAL: NCT06321783
Title: Investigation of the Relationship Between Cervical Proprioception and Cervical Muscle Endurance With Hand-eye Coordination and Postural Control in Individuals With Forward Head Posture
Brief Title: Relationship Between Cervical Proprioception and Endurance With Hand-eye Coordination and Postural Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Çoban, Research Assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-77082166-604.01.02-407303
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Forward Head Posture
Keywords: Forward Head Posture; Proprioception; Coordination; Postural Balance
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Other): Individuals with forward head posture
  Interventions: Other: Assessment
- Group 2 (Other): Individuals with normal head posture
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Evaluation of cervical proprioception, hand-eye coordination, postural control and endurance of cervical muscles

SUMMARY:
The aim of our study is to investigate the relationship between cervical proprioception and cervical muscle endurance with hand-eye coordination and postural control in individuals with forward head posture (FHP) and to compare them with a control group with normal head posture. After the demographic information and physical characteristics of the individuals are recorded, their craniovertebral angles (CVA) will be measured and they will be assigned to Group 1 (forward head posture) or Group 2 (normal head posture). Then, the individuals' cervical proprioception, hand-eye coordination, postural control and cervical muscle endurance values will be measured respectively. Cervical muscle endurance will be evaluated last, taking into account possible muscle fatigue, in order not to affect other measurement results. The recorded values will be compared between groups and the relationship of cervical proprioception and muscle endurance with hand-eye coordination and postural control will be examined. All evaluations will be made by the same researcher.

DETAILED DESCRIPTION:
Forward head posture is a malalignment defined as anterior translation of the head. This malalignment causes changes in cervical proprioception, decrease in the strength and endurance of the cervical muscles. A decrease in muscle endurance may cause a decrease in cervical proprioception. The cervical region is very important in terms of proprioceptive sensory input and has reflex connections to the (Central Nervous System) CNS. Therefore, abnormal proprioceptive sensory inputs received from cervical mechanoreceptors affect the CNS, which regulates postural control. It has been stated that FHP is associated with a decrease in static and dynamic balance. Head posture has an important role in the sensory information organization of the upper extremity. Hand-eye coordination allows the eyes to coordinate with hand movements.

Identifying the factors that may affect an individual with FHP is very important in planning the rehabilitation program.

The purpose of this study, investigate the relationship between cervical proprioception and cervical muscle endurance with hand-eye coordination and postural control in individuals with FHP and to compare them with a control group with normal head posture.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-24 years
* Volunteering to participate in the study

Exclusion Criteria:

* History of trauma or surgery involving the cervical or upper extremity
* Congenital anomaly of the cervical, thoracic or lumbar vertebra
* Abnormalities such as scoliosis
* Systemic arthritis or central nervous system disorders

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
Cervical Proprioception | Baseline
  Proprioception is the joint position sense. Cervical right and left rotation proprioception of individuals will evaluate with a digital inclinometer.
Hand-Eye Coordination | Baseline
  Individuals' hand-eye coordination will be evaluated by using the Alternate Wall Toss Test and recording the total number of times the ball is thrown and held against the wall without dropping it for 30 seconds.
Postural Stability Test | Baseline
  This test measures the participants' ability to keep the center of gravity within the limits of the support surface. Depending on the amount of deviation of the center of gravity from the center of the support surface, total stability index (TSI) scores will be recorded. The tests will be performed with eyes open and closed under the conditions of bipedal and unipedal (right side).
Stability Limit Test | Baseline
  In this test, which measures the dynamic balance control of the participants; movement and control skills are evaluated within the limits of the support surface of the center of gravity. Participants' percentage scores of the stability limit in all directions, total percentage score (overall) and time to complete the test (seconds) will be obtained.
Modified Sensory Organization Test | Baseline
  It evaluates the visual, somatosensory and vestibular sensory systems necessary for postural control.
  The test will be performed on firm and soft ground, with eyes open and closed conditions. At the end of the assessment, the sway index scores (SI-Sway Index) of all tested conditions will be obtained.
Endurance of Cervical Muscles | Baseline
  The endurance of the individuals' flexor and extensor muscles will be evaluated by recording the time in seconds that they can maintain the head position initially positioned by the therapist without changing it.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hazar, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MY, Lee HY, Yong MS. Characteristics of cervical position sense in subjects with forward head posture. J Phys Ther Sci. 2014 Nov;26(11):1741-3. doi: 10.1589/jpts.26.1741. Epub 2014 Nov 13. PMID 25435690
- [Background] Oliveira AC, Silva AG. Neck muscle endurance and head posture: A comparison between adolescents with and without neck pain. Man Ther. 2016 Apr;22:62-7. doi: 10.1016/j.math.2015.10.002. Epub 2015 Oct 22. PMID 26603679
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Background] Lee JH. Effects of forward head posture on static and dynamic balance control. J Phys Ther Sci. 2016 Jan;28(1):274-7. doi: 10.1589/jpts.28.274. Epub 2016 Jan 30. PMID 26957773